CLINICAL TRIAL: NCT03478085
Title: Near Infrared Spectroscopy-Guided Exercise Training in Peripheral Arterial Disease
Brief Title: Near-Infrared Spectroscopy-Guided Exercise Training in Peripheral Arterial Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13GRNT1693006
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional exercise therapy (Active Comparator): Training will be performed three times a week for 12 weeks. Each session will take place on a GaitKeeper treadmill (Sammons Preston, IL) treadmill and will last 45 minutes with a 5 minute warm up and cool down of either cycling or walking.
  Interventions: Other: Oxygen guided exercise therapy
- Oxygen guided exercise therapy (Experimental): Training will be performed three times a week for 12 weeks. Each session will take place on a GaitKeeper treadmill (Sammons Preston, IL) treadmill and will last 45 minutes with a 5 minute warm up and cool down of either cycling or walking. All patients will be outfitted during exercise with the PortaMon NIRS device on the most affected calf (including subjects in the symptom-driven exercise cohort). The intensity of training will be adjusted to either pain (claudication) rating or oxygen tension. In preliminary studies, a 50% reduction in the tissue saturation index is typically not associated with severe claudication and will be used as the lower level threshold to gauge physical effort (i.e., if subjects do not desaturate by >50% then the intensity of training - the walking pace - will be increased). The training duration, intensity, pain rating, and oxygen tension will be recorded.
  Interventions: Other: Oxygen guided exercise therapy
- Control (Placebo Comparator): Patients will be advised to walk independently.
  Interventions: Other: Oxygen guided exercise therapy

INTERVENTIONS:
Other: Oxygen guided exercise therapy — Subjects exercise to a certain intensity based on 15% muscle oxygen desaturation.

SUMMARY:
Background: Patients suffering with atherosclerotic peripheral arterial disease (PAD) have limited therapeutic options to improve claudication. Supervised exercise programs are generally effective in improving leg pain from walking, but are poorly adhered to because of patient discomfort. The benefit of exercise training programs is thought to be mediated in part through repeated ischemic stimuli that activate endogenous regenerative mechanisms. In preliminary studies, exercise-induced tissue desaturation by near infrared spectroscopy (NIRS) precedes the onset of leg pain. This proposal aims to explore a novel strategy of exercise training in PAD based on measured tissue hypoxia rather than pain symptoms using NIRS to non-invasively characterize muscle oxygen tension.

Methods: In subjects with symptomatic peripheral arterial disease, the efficacy of a novel NIRS-based strategy of thrice-weekly exercise training will be assessed. Enrolled subjects will be randomized to NIRS-based training, traditional claudication-based training, or self-directed walking. The hypotheses tested include: 1) NIRS-directed exercise improves claudication to a similar degree as symptom-directed exercise training and 2) is superior to self-directed walking. In the symptom-based group, physical effort will be dictated by claudication symptoms, whereas in the hypoxia-based training program, physical effort is dictated by NIRS measure of calf oxygen tension. Efficacy in the training programs will be evaluated by total walking time on a standard graded treadmill test after 12 weeks. Other measures will be claudication onset time, subjective and objective measures of physical activity, changes in vascular function. In addition, the hypothesis that hypoxia-directed training will result in increased ischemic signaling and increased progenitor cell mobilization to a degree similar as in claudication-based training will be tested.

Conclusions: These experiments will test whether a training strategy based on tissue hypoxia (measured by NIRS) is as effective as and more tolerable than traditional symptom-based training programs in PAD. In addition, these experiments will characterize mechanistic responses to hypoxia that may account for clinical improvements that exercise training affords.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Clinically stable symptoms of intermittent claudication from PAD (with no change in symptom severity in the 2 months prior to screening.)
* On stable medical therapy for previous 3 months.
* Able to achieve Total Walking Time (TWT) between 1 and 12 minutes on a standardized Gardner treadmill protocol.
* PAD will be defined by the presence of a Doppler-derived ankle-brachial index (ABI) of < 0.85 in the symptomatic limb after 10 minutes of rest at screening. For subjects with an ABI of >1.3 (non-compressible arteries) a Toe-Brachial Index (TBI) of < 0.70 must be obtained for subject qualification, or if ABI is > 0.85 to 1.0, and a reduction of 20% in ABI measured within 1 minute of treadmill testing.

Exclusion Criteria:

* Critical limb ischemia either chronic (category 3 and 4 of SVS classification) or acute ischemia manifested by rest pain, ulceration, or gangrene;
* Lower extremity vascular surgery, angioplasty or lumbar sympathectomy within 3 months of enrollment
* Unstable angina, myocardial infarction, transient ischemic attack, stroke or revascularization in the preceding 4 months;
* Severe heart failure (Class III or IV);
* Limitation on exercise for symptoms other than intermittent claudication such as arthritis or severe dyspnea;
* Alcohol or drug abuse, or any other disease process that, in the opinion of the PI, will interfere with the ability of the patient to participate in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Pain Free Walking Time in Minutes | 12 weeks
  Time until onset of claudication will be measured in subjects undergoing a Gardner protocol 12 minute walk on a treadmill.

SECONDARY OUTCOMES:
Total Treadmill Walking Time in Minutes | 12 weeks
  Time until onset of claudication will be measured in subjects undergoing a Gardner protocol 12 minute walk on a treadmill.

IPD SHARING:
Plan to Share IPD: No